CLINICAL TRIAL: NCT01515657
Title: A Randomized, Actively Controlled, Crossover Pharmacodynamic Evaluation of PL2200 Versus Enteric-Coated and Immediate Release Aspirin in Patients With Type II Diabetes
Brief Title: Pharmacodynamic Evaluation of PL2200 Versus Enteric-Coated and Immediate Release Aspirin in Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PL-ASA-004
Record Dates: First submitted 2012-01-13; First posted 2012-01-24 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PL2200 Aspirin Capsules (Experimental): Investigational drug arm; crossover design
  Interventions: Drug: PL2200 Aspirin Capsules
- Immediate-Release Aspirin Tablets (Active Comparator): Active comparator; crossover design
  Interventions: Drug: Immediate-Release Aspirin Tablets
- Enteric-coated aspirin caplets (Active Comparator): Active comparator; crossover design
  Interventions: Drug: Enteric-coated aspirin caplets

INTERVENTIONS:
Drug: PL2200 Aspirin Capsules — 325 mg aspirin; once per day for 3 days
  Arms: PL2200 Aspirin Capsules
Drug: Immediate-Release Aspirin Tablets — 325 mg aspirin; once per day for 3 days
  Arms: Immediate-Release Aspirin Tablets
Drug: Enteric-coated aspirin caplets — 325 mg aspirin; once per day for 3 days
  Arms: Enteric-coated aspirin caplets

SUMMARY:
This study will determine if aspirin from PL2200, an investigational product, gets into the blood stream as quickly as plain aspirin and enteric coated aspirin, and to test whether PL2200 is able to prevent blood clots as effectively as these other products, when administered to patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults 21-79
* Body mass index (BMI) of 30-40 kg/m2
* Non-insulin-dependent type-2 diabetics (as confirmed by hemoglobin A1c (HbA1c) of > 6.4% and/or fasting plasma glucose of >125 mg/dL or current anti-diabetic medication)
* AA-induced platelet aggregation response of >60% within 3 hours prior to initial dose of study drug administration

Exclusion Criteria:

* Contraindications to aspirin
* Previous history of vascular disease
* Patient requires insulin
* Use of non-steroidal anti-inflammatory drugs, anti-secretory agents, antacids, and salicylate-containing nutritional supplements within 2 weeks of randomization

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MedPace Clinical Pharmacology, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Bhatt DL, Grosser T, Dong JF, Logan D, Jeske W, Angiolillo DJ, Frelinger AL 3rd, Lei L, Liang J, Moore JE, Cryer B, Marathi U. Enteric Coating and Aspirin Nonresponsiveness in Patients With Type 2 Diabetes Mellitus. J Am Coll Cardiol. 2017 Feb 14;69(6):603-612. doi: 10.1016/j.jacc.2016.11.050. Epub 2017 Jan 11. PMID 28089180

RESULTS

PARTICIPANT FLOW:
Groups:
- PL2200 Aspirin First, Then IR Aspirin Tablets, Then EC Aspirin: First Intervention Period:
  PL2200 Aspirin Capsules: 325 mg aspirin; once per day for 3 days (after 2-week washout period)
  Second Intervention Period:
  IR (immediate-release) aspirin tablets: 325 mg aspirin; once per day for 3 days (after 2-week washout period)
  Third Intervention Period:
  EC (enteric coated) aspirin: 325 mg aspirin; once per day for 3 days
- IR Aspirin Tablets First, Then EC Aspirin, Then PL2200 Aspirin: First Intervention Period:
  IR (immediate-release) aspirin tablets: 325 mg aspirin; once per day for 3 days (after 2-week washout period)
  Second Intervention Period:
  EC (enteric coated) aspirin: 325 mg aspirin; once per day for 3 days (after 2-week washout period)
  Third Intervention Period:
  PL2200 Aspirin Capsules: 325 mg aspirin; once per day for 3 days
- EC Aspirin First, Then PL2200 Aspirin, Then IR Aspirin Tablets: First Intervention Period:
  EC (enteric coated) aspirin: 325 mg aspirin; once per day for 3 days (after 2-week washout period)
  Second Intervention Period:
  PL2200 Aspirin Capsules: 325 mg aspirin; once per day for 3 days (after 2-week washout period)
  Third Intervention Period:
  IR (immediate-release) aspirin tablets: 325 mg aspirin; once per day for 3 days
Period: First Intervention
Arm/Group | PL2200 Aspirin First, Then IR Aspirin Tablets, Then EC Aspirin | IR Aspirin Tablets First, Then EC Aspirin, Then PL2200 Aspirin | EC Aspirin First, Then PL2200 Aspirin, Then IR Aspirin Tablets
Started | 14 | 13 | 13
Completed | 14 | 12 | 13
Not Completed | 0 | 1 | 0
Period: Second Intervention
Arm/Group | PL2200 Aspirin First, Then IR Aspirin Tablets, Then EC Aspirin | IR Aspirin Tablets First, Then EC Aspirin, Then PL2200 Aspirin | EC Aspirin First, Then PL2200 Aspirin, Then IR Aspirin Tablets
Started | 14 | 12 | 13
Completed | 14 | 11 | 13
Not Completed | 0 | 1 | 0
Period: Third Intervention
Arm/Group | PL2200 Aspirin First, Then IR Aspirin Tablets, Then EC Aspirin | IR Aspirin Tablets First, Then EC Aspirin, Then PL2200 Aspirin | EC Aspirin First, Then PL2200 Aspirin, Then IR Aspirin Tablets
Started | 14 | 11 | 13
Completed | 13 | 11 | 13
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All patients that received at least 1 dose of study drug under the study protocol.
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to 99% Inhibition of Serum Thromboxane (TxB2)
Description: Aspirin's antiplatelet activity is measured by the capacity of platelets to generate serum thromboxane (a surrogate marker for inhibition of COX-1 by aspirin). Inhibition of serum thromboxane is a key marker of antiplatelet efficacy.
Time Frame: 4 days
Population: Pharmacodynamic (PD) Evaluable Population for Time to 99% Inhibition
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PL2200 Aspirin Capsules | Immediate-Release Aspirin Tablets | Enteric-coated Aspirin Caplets
Number analyzed (Participants) | 35 | 35 | 35
Hours | 12.36 (23.42) | 16.65 (27.21) | 48.64 (31.20)

ADVERSE EVENTS:
Description: modified Intent-to-Treat population: all patients that received at least 1 dose of study drug under the study protocol
Arm/Group | PL2200 Aspirin Capsules | Immediate-Release Aspirin Tablets | Enteric-coated Aspirin Caplets
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 2/38 | 4/40 | 7/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PL2200 Aspirin Capsules (N=38) | Immediate-Release Aspirin Tablets (N=40) | Enteric-coated Aspirin Caplets (N=38)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Standard confidentiality agreement